CLINICAL TRIAL: NCT03716934
Title: CRyoAblation vs AntiaRrhythmic Drugs for Persistent Atrial Fibrillation Trial
Acronym: craft
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Nicasio Perez Castellano, Principal Investigator, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17/507-R_M
Record Dates: First submitted 2018-10-15; First posted 2018-10-23 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cryoablation (Experimental): Cryoablation for bidirectional block of all pulmonary veins
  Interventions: Device: Arctic Front Advance® balloon catheter; Device: Confirm RX heart monitor® (Abbott)
- Antiarrythmics (Active Comparator): The drug will be chosen based on the preference of the researcher based on clinical practice guidelines.
  Interventions: Drug: Antiarrhythmic drug; Device: Confirm RX heart monitor® (Abbott)

INTERVENTIONS:
Device: Arctic Front Advance® balloon catheter — Cryoablation of bidirectional block of all pulmonary veins
  Arms: Cryoablation
Drug: Antiarrhythmic drug — The drug will be chosen based on the preference of the researcher / responsible physician and current clinical practice guidelines.
  Other Names: Class I or III
  Arms: Antiarrythmics
Device: Confirm RX heart monitor® (Abbott) — Is a subcutaneous implantable device that provides continuous monitoring of the heart rate for more than 3 years without any effect on cardiac function

SUMMARY:
This is a prospective, randomized, multicenter study comparing the relative efficacy and safety of cryoablation of PVs using the Arctic Front Advance® balloon catheter with antiarrhythmic therapy in patients with persistent AF.

DETAILED DESCRIPTION:
The ablation of pulmonary veins is a very effective treatment for the treatment of paroxysmal atrial fibrillation. The benefit of the isolation of pulmonary veins in persistent atrial fibrillation seems to be minor and the level of scientific evidence available requires additional clinical trials to define the value of ablation in this type of patients.

The symptomatology of atrial fibrillation recurrences is variable among patients and among differens moments in the same patient. Pharmacological treatment and ablation have been used to reduce the symptomatology of atrial fibrillation recurrences and to increase the proportion of asymptomatic recurrences. Different forms of electrical monitoring of the heart rate are used to evaluate the effectiveness of an intervention. Frequents monitoring periods provide the information of the heart rate and the effect of any intervention.

The "Confirm RX heart monitor® (Abbott)" is a subcutaneous implantable device that provides continuous monitoring of the heart rate for more than 3 years without any effect on cardiac function. This implantable Holter automatically detects and saves atrial and ventricular arrhythmic episodes. The device can be analyzed in person or remotely, and can help to make decisions regarding anticoagulant and antiarrhythmic treatment of patients, while representing a powerful research tool for evaluate the effectiveness of different therapeutic options.

This is a prospective, randomized, multicenter study that compares the relative efficacy and safety of cryoablation of pulmonary veins using the Arctic Front Advance® balloon catheter with antiarrhythmic treatment in patients with persistent atrial fibrilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent persistent atrial fibrilation

Exclusion Criteria:

* Patients with atrial fibrilation for more than one year at baseline
* Atrial fibrilation prior ablation
* Age> 75 years or <18 years
* Hyperthyroidism
* Hypertrophic cardiomyopathy
* Severe valvular disease (stenosis or regurgitation)
* Carriers of cardiac valves
* Anteroposterior diameter of left atrium> 50 mm (left parasternal long axis)
* Contraindications for anticoagulation
* Left atrial thrombus
* Anemia
* Active infection
* Pregnancy
* Atrial fibrilation secondary to transient, avoidable or correctable causes (hyperthyroidism, pneumonia, pulmonary embolism, drugs, hydroelectrolytic alterations ...)
* Life expectancy of less than 24 months
* Participation in another non-purely observational study
* Patients unable to understand treatment and / or study and / or providing adequate informed consent
* Any condition, that in the opinion of the physician responsible for the patient, contraindicates any of the treatments of the study
* Microalbuminemia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

PRIMARY OUTCOMES:
Survival time with atrial fibrilation, auricular flutter or tachycardia | Up to 9 months.
  Survival time without atrial fibrilation, atrial flutter or atrial tachycardia of more than 2 minutes duration detected by Holter
Presence of death or one major complications. | first month
  Presence of death or one of the following major complications: Stroke, systemic embolism, acute myocardial infarction, cardiac tamponade, need for transfusion, diaphragmatic paralysis lasting more than 24 hours or causing respiratory failure, atrioesophageal fistula, stenosis of pulmonary veins, Sustained (> 30 sec) or symptomatic ventricular tachycardia, Syncope secondary to bradyarrhythmias or tachyarrhythmias, Need for hospitalization due to cardiovascular causes or related to the study treatments, Any Serious Adverse Reaction or Serious Adverse Event related to the study treatments.
Presence of death or one major complications. | fourth month
  Presence of death or one of the following major complications: Stroke, systemic embolism, acute myocardial infarction, cardiac tamponade, need for transfusion, diaphragmatic paralysis lasting more than 24 hours or causing respiratory failure, atrioesophageal fistula, stenosis of pulmonary veins, Sustained (> 30 sec) or symptomatic ventricular tachycardia, Syncope secondary to bradyarrhythmias or tachyarrhythmias, Need for hospitalization due to cardiovascular causes or related to the study treatments, Any Serious Adverse Reaction or Serious Adverse Event related to the study treatments.
Presence of death or one major complications. | thirteen month
  Presence of death or one of the following major complications: Stroke, systemic embolism, acute myocardial infarction, cardiac tamponade, need for transfusion, diaphragmatic paralysis lasting more than 24 hours or causing respiratory failure, atrioesophageal fistula, stenosis of VP, Sustained (> 30 sec) or symptomatic ventricular tachycardia, Syncope secondary to bradyarrhythmias or tachyarrhythmias, Need for hospitalization due to cardiovascular causes or related to the study treatments, Any Serious Adverse Reaction or Serious Adverse Event related to the study treatments.

SECONDARY OUTCOMES:
Percentage of patients without atrial fibrilation, flutter or tachycardia | first month
  Number of patients without atrial fibrilation, atrial flutter or atrial tachycardia of more than 2 minutes
Percentage of patients without atrial fibrilation, flutter or tachycardia | fourth month
  Number of patients without atrial fibrilation, atrial flutter or atrial tachycardia of more than 2 minutes
Percentage of patients without atrial fibrilation, flutter or tachycardia | thirteen month
  Number of patients without atrial fibrilation, atrial flutter or atrial tachycardia of more than 2 minutes
Percentage of patient with cardioversion | first month
  Number of patients that need cardioversion
Percentage of patient with cardioversion | fourth month
  Number of patients that need cardioversion
Percentage of patient with cardioversion | thirteen month
  Number of patients that need cardioversion
Percentage of patient with need to consult the emergency room or hospitalization due to cardiovascular events | first month
  Number of patients that need to consult the emergency room or hospitalization due to cardiovascular events
Percentage of patient with need to consult the emergency room or hospitalization due to cardiovascular events | fourth month
  Number of patients that need to consult the emergency room or hospitalization due to cardiovascular events
Percentage of patient with need to consult the emergency room or hospitalization due to cardiovascular events | thirteen month
  Number of patients that need to consult the emergency room or hospitalization due to cardiovascular events
Percentage of patient with need a change or suspension of antiarrhythmic due to inefficiency | first month
  Number of patients that need a change or suspension of antiarrhythmic due to inefficiency
Percentage of patient with need a change or suspension of antiarrhythmic due to inefficiency | fourth month
  Number of patients that need a change or suspension of antiarrhythmic due to inefficiency
Percentage of patient with need a change or suspension of antiarrhythmic due to inefficiency | thirteen month
  Number of patients that need a change or suspension of antiarrhythmic due to inefficiency
Percentage of patient with need for ablation or re-ablation not scheduled | first month
  Number of patients that need a ablation or re-ablation not scheduled
Percentage of patient with need for ablation or re-ablation not scheduled | fourth month
  Number of patients that need a ablation or re-ablation not scheduled
Percentage of patient with need for ablation or re-ablation not scheduled | thirteen month
  Number of patients that need a ablation or re-ablation not scheduled

CONTACTS AND LOCATIONS:
Locations (1):
- Fundacion para Investigación Biomedica Hospital Clinico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No